CLINICAL TRIAL: NCT06863376
Title: Evaluating the Safety and Efficacy of Carbocisteine in the Treatment of Nonalcoholic Fatty Liver Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1478
Record Dates: First submitted 2025-03-01; First posted 2025-03-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Carbocysteine; Exercise; Walking

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients will receive the standard conventional therapy in addition to placebo for 3 months.
  Interventions: Other: Physical activity, walking, and calorie restriction
- Carbocistiene group (Active Comparator): Patients will be given the standard conventional therapy plus carbocistiene 375 mg two times daily.
  Interventions: Drug: Carbocysteine 375 MG; Other: Physical activity, walking, and calorie restriction

INTERVENTIONS:
Drug: Carbocysteine 375 MG — Carbocysteine is a muco-active drug with free radical scavenging and anti-inflammatory properties. It is actually approved for clinical use as adjunctive therapy of respiratory tract disorders
  Arms: Carbocistiene group
Other: Physical activity, walking, and calorie restriction — • The standard conventional therapy in both groups included regular exercise in the form of any physical activity as walking, cycling, etc. for 30-45 minutes minimum 5 days per week in addition to calorie restriction in overweight and obese patients

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a global public health concern, and the leading cause of chronic liver disease, especially in developed countries. NAFLD is characterized by lipid accumulation in the liver not attributed to other causes. Lifestyle interventions, including dietary modification and exercise, remain the cornerstone of NAFLD treatment. Pharmacological treatments aimed primarily at improving liver disease should generally be limited to those with biopsy-proven NASH and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Either male or female adult patients (>18 years) with fatty liver diagnosis by using upper abdominal ultrasound echography

Exclusion Criteria:

* Pregnant and/or lactating women
* Excessive alcohol use (defined as an average alcohol intake > 30 g per day in men and > 20 g per day in women)
* Other etiology of chronic liver diseases such as viral hepatitis, drug-induced hepatitis, autoimmune hepatitis.
* patients suffering from chronic kidney disease, and hyper/hypoparathyroidism
* Hypersensitivity to carbocistiene.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
The change in the degree of steatosis in the Ultra Sound | 3 months
  The change in the degree of steatosis in the Ultra Sound

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt